CLINICAL TRIAL: NCT01204697
Title: A Randomized Phase II Trial of Erlotinib or Intermittent Dosing of Erlotinib and Docetaxel in Male Former-smokers With Locally Advanced or Metastatic Squamous NSCLC in Second-line Setting After Failure on Chemotherapy
Brief Title: A Study of Erlotinib [Tarceva] as Monotherapy or Intermittent Dosing With Docetaxel in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer. (TALISMAN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21869
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Results first posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Docetaxel; Erlotinib Hydrochloride

ARMS (2):
- A (Experimental)
  Interventions: Drug: erlotinib [Tarceva]
- B (Experimental)
  Interventions: Drug: docetaxel; Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: docetaxel — 75 mg/m2 intravenously every 3 weeks for 4 cycles
  Arms: B
Drug: erlotinib [Tarceva] — 150 mg/day orally, days 2-16 each 3-week cycle for 4 cycles; 150 mg/day orally thereafter
  Arms: B
Drug: erlotinib [Tarceva] — 150 mg/day orally as monotherapy
  Arms: A

SUMMARY:
This randomized parallel group study will assess the efficacy and safety of erlotinib [Tarceva], as monotherapy or intermittent dosing with docetaxel, in second-line setting in former-smoker male patients with advanced or metastatic squamous non-small cell lung cancer. Patients will be randomized to receive either Tarceva (150 mg/day orally) as monotherapy or 4 cycles of docetaxel (75 mg/m2 intravenously every 3 weeks) plus Tarceva (150 mg/day orally, days 2-16 each cycle) followed by Tarceva monotherapy. Anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* male patients, >/=18 years of age
* former smoker (smoked >/= 100 cigarettes in his lifetime and quit >12 months before enrollment)
* locally advanced (stage IIIb), metastatic (stage IV) or recurrent squamous non-small cell lung cancer
* prior platinum-based therapy for advanced NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* uncontrolled symptomatic central nervous system (CNS) metastases
* prior therapy against epidermal growth factor receptor (EGFR)
* >1 prior chemotherapy for advanced/metastatic NSCLC
* radiotherapy <28 days prior to enrollment
* history of melanoma at any time, or another malignancy in the last 5 years except for carcinoma in situ of the cervix, basal or squamous cell carcinoma of the skin, or surgically cured malignant neoplasias with a disease-free interval of >5 years
* not fully treated eye inflammation or infection, or predisposing conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Italy (18):
  - Lecce, Apulia
  - San Giovanni Rotondo, Apulia
  - Avellino, Campania
  - Napoli, Campania
  - Parma, Emilia-Romagna
  - Aviano (PN), Friuli Venezia Giulia
  - Rome, Lazio
  - Cremona, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Pavia, Lombardy
  - Sondalo, Lombardy
  - Macerata, The Marches
  - Lido di Camaiore, Tuscany
  - Pisa, Tuscany
  - Pontedera, Tuscany
  - Treviso, Veneto
  - Vicenza, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Participants received erlotinib (Tarceva) at a dose of 150 milligram per day (mg/day) orally as monotherapy, up to progressive disease (PD), death, or unacceptable toxicity.
- Docetaxel and Erlotinib: Participants received docetaxel at a dose of 75 milligram per square meter (mg/m^2) as an intravenous infusion on Day 1 of each 3-week cycle, and erlotinib at a dose of 150 mg/day orally from Day 2 to Day 16 of each 3-week cycle for 4 cycles, administered in absence of PD, death, or unacceptable toxicity. Following the 4 cycles, erlotinib 150 mg/day was administered orally as monotherapy up to PD, death or unacceptable toxicity.
Period: Overall Study
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Started | 36 | 38
Treated | 36 | 37
Completed | 5 | 2
Not Completed | 31 | 36
Not completed — Death | 26 | 27
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Randomized, but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received at least one dose of study medication. Participants were analyzed according to treatment received.
Groups:
- Erlotinib: Participants received erlotinib at a dose of 150 mg/day orally as monotherapy, up to PD, death, or unacceptable toxicity.
- Docetaxel and Erlotinib: Participants received docetaxel at a dose of 75 mg/m^2 as an intravenous infusion on Day 1 of each 3-week cycle, and erlotinib at a dose of 150 mg/day orally from Day 2 to Day 16 of each 3-week cycle for 4 cycles, administered in absence of PD, death, or unacceptable toxicity. Following the 4 cycles, erlotinib 150 mg/day was administered orally as monotherapy up to PD, death or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Docetaxel and Erlotinib | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.3) | 65.9 (8.1) | 67.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free From Disease Progression or Death at 6 Months
Description: According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, progressive Disease (PD) is defined as: for Target Lesions - At least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). (Note: the appearance of one or more new lesions is also considered progression). For Non-Target Lesions - Unequivocal progression of existing non-target lesions. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Month 6
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Number analyzed (Participants) | 36 | 37
percentage of participants | 8.3 [0.0 to 17.4] | 8.1 [0.0 to 16.9]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free Survival (PFS) was defined as the interval (in days) between the date of randomization and the first documentation of progressive disease or death from any cause. Participants alive and progression-free were considered as censored at the date of the last tumor assessment when the participant was known to be progression-free. Participants without post-baseline tumor assessment, but known to be alive, were censored at the time of randomization. PFS (days) = (Date of Event - Date of Randomization) + 1. PFS was assessed using the Kaplan-Meier method. Detailed definition of PD is provided in Outcome Measure 1.
Time Frame: From randomization until progressive disease or death, assessed up to 18 months
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Number analyzed (Participants) | 36 | 37
months | 2.33 [2.13 to 4.13] | 2.82 [2.30 to 3.97]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the interval (in days) between the date of randomization and death from any cause. Participants alive at the time of the analysis were censored at the date they were last known to be alive. OS was assessed using the Kaplan-Meier method.
Time Frame: From randomization until death, assessed up to 18 months
Population: FAS population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Number analyzed (Participants) | 36 | 37
months | 5.61 [3.54 to 8.69] | 8.95 [6.13 to 10.4]

4. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Best overall response (complete response [CR]/partial response [PR]) was defined as the best response recorded from the start of the treatment until disease progression (PD). Best response in this trial was defined as the best response observed at any post-treatment visits. According to RECIST Version 1.1, CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 mm). No new lesions. PR was defined as greater than or equal to [>=] 30% decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: From randomization until progressive disease or death, assessed up to 18 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Number analyzed (Participants) | 36 | 37
percentage of participants | 2.8 [0.0 to 8.15] | 8.1 [0.0 to 16.9]

5. Secondary Outcome: Percentage of Participants With Disease Control
Description: Disease control was defined as PR, CR, or SD. Participants who did not achieve a CR or PR or SD were counted as non-responders in the analysis of disease control. According to RECIST Version 1.1, SD was defined as not qualifying for CR, PR, and PD. Detailed definitions of CR and PR are provided in Outcome Measure 4.
Time Frame: From randomization until progressive disease or death, assessed up to 18 months
Population: FAS population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Number analyzed (Participants) | 36 | 37
percentage of participants | 41.7 [25.6 to 57.8] | 37.8 [22.2 to 53.5]

6. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response (DoR) was defined as the interval (in days) from first documentation of a response (CR/PR depending on which occurred first) to the date of the first documentation of disease progression or death from any cause. Participants presenting a response were considered as censored at the date of the last assessment with a documentation of non-progression. DoR (days) = (Date of PD/death - Date of CR/PR) + 1. Assessments were performed according to RECIST Version 1.1. DoR was assessed using the Kaplan-Meier method. Detailed definitions of CR and PR are provided in Outcome Measure 4.
Time Frame: From randomization until progressive disease or death, assessed up to 18 months
Population: FAS population. Here, number of participants analyzed signifies those participants who had a best overall response of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Number analyzed (Participants) | 1 | 3
months | NA [NA to NA] — Median and corresponding 95% confidence interval were not estimable as the only participant evaluable was censored. | 8.69 [1.87 to 10.8]

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | Erlotinib | Docetaxel and Erlotinib
Serious Adverse Events (participants affected / at risk) | 15/36 | 10/37
Other Adverse Events (participants affected / at risk) | 32/36 | 35/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=36) | Docetaxel and Erlotinib (N=37)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Device dislocation (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Performance status decreased (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Uncoded (General disorders) | 0 | 1
Angiopathy (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=36) | Docetaxel and Erlotinib (N=37)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 9
Tachycardia (Cardiac disorders) | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 14
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 5
Asthenia (General disorders) | 8 | 10
Chest pain (General disorders) | 5 | 0
Mucosal inflammation (General disorders) | 0 | 5
Pyrexia (General disorders) | 4 | 6
Hypertransaminasaemia (Hepatobiliary disorders) | 3 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 2
Folliculitis (Infections and infestations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Coordination abnormal (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 16 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.